CLINICAL TRIAL: NCT00519051
Title: Efectividad de la Farmacoterapia Monitorizada en Pacientes Deprimidas de la atención Primaria de Salud y su repercusión Sobre la Salud Mental de Sus Hijos
Brief Title: A Randomized Clinical Trial for Depressed Mothers at Primary Care Level
Acronym: DMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1040432
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Depression
Keywords: depression; primary care; pharmacotherapy
MeSH Terms: conditions — Depression | interventions — Antidepressive Agents; Fluoxetine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- control group (Active Comparator): patients can receive pharmacotherapy and psychotherapy and specialized treatment
  Interventions: Other: monitorized pharmacotherapy with antidepressants drugs (Fluoxetine)

INTERVENTIONS:
Other: monitorized pharmacotherapy with antidepressants drugs (Fluoxetine) — Fluoxetine oral,20-60 mg/day for 6 months with telephone monitorization
  Other Names: usual care

SUMMARY:
A randomized clinical trial was carried out at primary care level in Santiago, Chile to compare a pharmacological intervention for depressed mothers controlled by phone from a central level (TM) and the usual treatment (TH) and its impact on children's mental health.

Hypothesis: pharmacological intervention for depression controlled by phone from a central level will be more effective than usual care in depressed mothers.

DETAILED DESCRIPTION:
Aim:to compare a pharmacological intervention for depressed mothers controlled by phone from a central level (TM) and the usual treatment (TH) and its impact on children's mental health.

Material and methods: A RCT wasw carried out at primary care clinics in Santiago.Sample:three hundred and forty five depressed women . One children of each mother was randomly selected. Women are randomly assigned to receive the usual therapy or a pharmacological intervention with periodical telephone contacts with medical collaboration personnel, to reinforce compliance with treatment and educate about the disease, for 6 months. Women were blindly evaluated at 3, 6 and 12 months with the Hamilton depression rating score (HDRS) and the SF-36 to assess depressive symptoms and quality of life, respectively; the Dyadic Adjustment Scale to assess marital adjustment.

Child psychopathology was assessed with the Child Behavior Checklist (CBCL), the Brief Psychiatric Rating Scale for Children (BPRS-C), Screen for Child Anxiety Related Emotional Disorders(SCARED)and the Children's Depression Inventory.

ELIGIBILITY:
Inclusion Criteria:

* depressed mothers with al least one child aged 6-16

Exclusion Criteria:

* currently treatment for depression,psychosis,bipolar depression,alcohol or drug abuse, gravidity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2004-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
depressive symptoms measured with the HDRS | at 3,6 and 12 months after randomization

SECONDARY OUTCOMES:
quality of life measured with the SF-36 | at 3,6 and 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: rosemarie fritsch, MD, Principal Investigator — University of Chile
Locations (1):
- CORESAM Conchali, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Result] Fritsch R, Araya R, Solis J, Montt E, Pilowsky D, Rojas G. [A randomized trial of pharmacotherapy with telephone monitoring to improve treatment of depression in primary care in Santiago, Chile]. Rev Med Chil. 2007 May;135(5):587-95. Epub 2007 Jul 9. Spanish. PMID 17657327